CLINICAL TRIAL: NCT01726647
Title: Metabolism Associated With Abdominal Fat Mass Distribution
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: 08.02.NRC
Record Dates: First submitted 2012-11-06; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Obese
Keywords: obese women; fat mass distribution; Metabolomic profiles
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No product is tested: No intervention

SUMMARY:
Objectives:

The primary objective of this clinical trial is to characterize metabolic signatures associated with abdominal fat distribution in 40 women with different BMI 29-40 and different abdominal distribution of fat (visceral vs. sub-cutaneous fat).

No intervention with a product is planned. The subjects will be given one high fat meal with commercial products (eggs, milk, cream, bread, fruits, cheese and cheese) on one test day to test the post-prandial metabolic response.

ELIGIBILITY:
Inclusion Criteria:

* BMI 29-40 kg/m2
* Aged 25-45

Exclusion Criteria:

* Diagnosed metabolic disorder such as Diabetes type 1 and 2, cardiovascular disease, metabolic syndrome
* Pregnancy
* Any pathology (infectious or other) having required an antibiotic therapy within 1 month prior to the beginning of the study.
* Any therapy (contraception apart) within the run-in period of one week before the test day.
* Subject who cannot be expected to comply with treatments and measures.
* Subject who is affected by any specific eating disorder
* Currently participating or having participated in another clinical trial during the last 3 months prior to the beginning of this study.
* Subjects having recently undergone a weight loss of more than 3 kilos during the last 3 months

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Obese women
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Metabolic plasma, urine and faeces profiles as a function of fat mass distribution | Changes from baseline in metabolic profiles at one day following fat meal intake
  Metabolic profiles of plasma, urine and feces samples are obtained by Nuclear Magnetic Resonance spectroscopy and Mass Spectrometry.
  Fat mass distribution is assessed using CT scan and DXA (Dual X-Ray Energy Absorptiometry).

SECONDARY OUTCOMES:
Insulin sensitivity | Measured on the day before the fat meal intake
  Insulin sensitivity is measured by oral glucose tolerance test
Basal Energy Expenditure | Basal Energy Expenditure is measured on the day preceding the fat meal intake
  Basal Energy Expenditure is measured by indirect calorimetry

CONTACTS AND LOCATIONS:
Overall Officials: Vittorio Giusti, MD, PD/MER, Principal Investigator — University Hospitals of Lausanne
Locations (2):
- Switzerland (2):
  - Nestlé Clinical Development Unit / Metabolic Unit, Lausanne
  - University Hospitals, Service of endocrinology, diabetology, and metabolism, Lausanne